CLINICAL TRIAL: NCT01755845
Title: Phase III Randomized Study of Concurrent Paclitaxel/Cisplatin Chemotherapy and Radiotherapy With or Without Consolidation Chemotherapy in High-Risk Patients With Early-Stage Cervical Cancer Following Radical Hysterectomy
Brief Title: Trial of Postoperative Chemoradiotherapy With or Without Consolidation Chemotherapy for Cervical Cancer Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: xie congying (Other)
Responsible Party: Sponsor-Investigator, xie congying, Director, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WZMC-11256
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; radiotherapy; postoperative therapy; chemotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Paclitaxel; Cisplatin; Radiotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Patients in this arm will postoperatively receive paclitaxel 135 mg/m2 d1 and cisplatin 25mg/m2 d1-3 intravenously every 4 weeks with radiation. Radiotherapy consisted of 46-50 gray (5 x 2.0 gray/week) on pelvic area. After completion of chemoradiotherapy, patients receive paclitaxel 135 mg/m2 d1 and cisplatin 25mg/m2 d1-3. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: paclitaxel; Drug: cisplatin; Radiation: radiotherapy
- Arm 2 (Active Comparator): Patients receive chemoradiotherapy as in arm 1.
  Interventions: Drug: paclitaxel; Drug: cisplatin; Radiation: radiotherapy

INTERVENTIONS:
Drug: paclitaxel
Drug: cisplatin
Radiation: radiotherapy

SUMMARY:
The purpose of this study is to determine the efficacy and safety of consolidation chemotherapy with paclitaxel plus cisplatin (2 cycles per 3 weeks) following radical hysterectomy and adjuvant chemoradiation (2 cycles per 4 weeks) for high risk early stage cervical cancer.

DETAILED DESCRIPTION:
Cervical carcinoma is one of the most common gynecologic cancers worldwide. Early stage cervical cancer can be treated effectively with either radiotherapy or radical hysterectomy plus pelvic lymph node dissection. However, several pathological risk factors, such as lymph node metastasis, the involvement of vaginal resection margin, and the parametrial invasion, have been identified to compromise the patient prognosis.

Concurrent radiotherapy with cisplatin-based chemotherapy has become the standard treatment for patients with cervical cancer. However, many patients with pathological risk factors treated with concurrent radiotherapy plus single agent cisplatin still suffered from the local or distant relapse. How to improve the treatment outcome of these patients is a very important issue and requires further clinical investigation.

Paclitaxel has been demonstrated to be a good radiosensitizer. In addition, paclitaxel/cisplatin combination chemotherapy was demonstrated to have superior progression-free survival than platinum alone in some phase Ⅱ studies. In addition, it is not yet known whether chemotherapy and radiation therapy are more effective when given with consolidation chemotherapy in treating cervical cancer.

Therefore, the investigators are going to perform the efficacy and safety study of postoperative concurrent paclitaxel/cisplatin chemotherapy and radiotherapy with consolidation chemotherapy in high-risk patients with early-stage cervical cancer following radical hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Undertaken radical hysterectomy with diagnosis of invasive cervical cancer I a2-II b (non-small cell type)
* One or more risk factors (lymph node involvement, resection margin involvement, parametrial involvement)
* Eastern Cooperative Oncology Group 0-2
* Expected life span over 6 months.
* No distant metastasis
* Adequate bone marrow functions (absolute neutrophil count≥ 1,500/ul, blood platelet≥ 100,000/ul, haemoglobin≥ 10g/dl)
* Adequate renal functions(serum creatinine ≤ 1.5mg/dl)
* Adequate liver functions (serum bilirubin ≤ 1.5mg/dl, aspartate aminotransferase/alanine aminotransferase ≤ 3 times(normal value)
* Written informed consent

Exclusion Criteria:

* Previous history of chemotherapy or radiation
* Hypersensitive reaction to platinum/paclitaxel agent
* History of other cancer
* Concurrent systemic illness not appropriate for chemotherapy
* Active infection requiring antibiotics
* Pregnancy
* Metastasis to paraaortic lymph node

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 3 years

SECONDARY OUTCOMES:
overall survival | 5 years

OTHER OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | 1 year
  assessed by NCI Common Terminology Criteria v3.0

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China